CLINICAL TRIAL: NCT04534140
Title: Evaluating the Effect of an Antioxidant Nutraceutical on Skin Health, as Measured by Investigator Global Assessment, Quality-of-Life, and Corneometry, in Persons With Mild to Moderately Severe Facial Acne Vulgaris
Brief Title: Skin Hydration in Persons With Acne After Dietary Supplementation With Botanical Antioxidants
Acronym: KIWIBOOSTER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Contract not negotiated.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19-002095
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Acne Vulgaris; Acne
Keywords: antioxidants; acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: This will be a 2-armed investigational group (botanical dietary supplement) and placebo group (supplement vehicle), double-blind, randomized, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBKB Capsule (Experimental): Experimental group participants will take one capsule of the HBKB botanical dietary supplement orally, once daily
  Interventions: Dietary Supplement: HBKB Capsule
- HBKB Capsule Vehicle (Placebo Comparator): Control group participants will take one capsule of the HBKB botanical dietary supplement vehicle orally, once daily
  Interventions: Other: HBKB Supplement Vehicle

INTERVENTIONS:
Dietary Supplement: HBKB Capsule — The botanical dietary supplement 'Halo Beauty Kiwi Booster' (HBKB) taken daily orally.
  Arms: HBKB Capsule
Other: HBKB Supplement Vehicle — Control group participants will take one capsule of the HBKB botanical dietary supplement vehicle orally, once daily
  Arms: HBKB Capsule Vehicle

SUMMARY:
Antioxidants have been studied for their abilities to combat reactive oxygen species in a multitude of conditions. This study aims to assess whether the botanical dietary supplement 'Halo Beauty Kiwi Booster' (HBKB), taken orally daily for 8 weeks, can assist with Acne vulgaris as well as skin hydration and quality of life for those with acne.

DETAILED DESCRIPTION:
The study will be a 2-armed investigational trial with one group receiving botanical dietary supplement and one placebo group provided with the similar supplement vehicle. The trial will be double-blind, randomized, parallel-group study. The investigational group will receive the botanical dietary supplement 'Halo Beauty Kiwi Booster' (HBKB), to be taken orally daily for 8 weeks. Control group participants will receive the HBKB botanical dietary supplement vehicle as a placebo to be taken orally daily for 8 weeks.Participants will have their skin assessed

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-35 years of age able to provide consent to participate
* IGA of mild to moderately severe facial Acne Vulgaris (AV) at screening
* Potential participants with mild to moderately severe facial AV and with AV on their neck, shoulders, chest and/or back body surface areas may be included.

Exclusion Criteria:

* An Investigator Global Assessment IGA of severe facial, neck, back or truncal AV
* Diagnosis of a chronic inflammatory disease such as lupus, multiple sclerosis, cancer, Chron's disease or cancer
* Allergies to Astaxanthin (microalgae), Grape Seed Extract, Kiwi fruit or Kiwi extract, Pineapple fruit or extract (bromelain), Rosehip or Rosehip extract, Gooseberry, Rosehip, Grapes
* Secondary AV, such as occupational AV, steroid induced AV, or AV associated with endocrine disorders
* Having facial dermatosis that may interfere evaluations by IGA such as sunburn, eczema, psoriasis, erythematotelangectatic rosacea or seborrheic dermatitis
* Use of isotretinoin within 2 months
* Use of adapalene or tretinoin within 2 weeks
* Use of anti-biotics within 2 weeks
* Use of oral corticosteroids or androgens within 2 weeks
* Use of anticonvulsants
* Any subject who the PI deems unsuitable for any reason

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2023-01-24 (Estimated); Study Completion 2023-01-24 (Estimated)

PRIMARY OUTCOMES:
Botanical Impact on hydration in those with Acne Vulgaris | 8 weeks
  To prospectively appraise changes in stratum corneum hydration levels in persons with Acne Vulgaris (AV) after dietary supplementation with a compilation of botanical antioxidants.

SECONDARY OUTCOMES:
Botanical Impact on Acne Vulgaris | 8 weeks
  To prospectively appraise changes in Investigator Global Assessment (IGA) of Facial AV after dietary supplementation with a compilation of botanical antioxidants.Scale is 0-4 (0 - clear and 4 - severe)
Botanical Impact on Quality of Life in those with Acne | 8 weeks
  To prospectively appraise changes in AV related quality-of-life (AVQoL) after dietary supplementation with a compilation of botanical antioxidants.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, Principal Investigator — UCLA Professor of Medicine
Locations (1):
- UCLA Center for Human Nutrition, 1000 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No